CLINICAL TRIAL: NCT00068159
Title: Characterization of Cardiac Function in Subjects With Hereditary Hemochromatosis Who Are New York Heart Association Functional Class I
Brief Title: Cardiac Function in Patients With Hereditary Hemochromatosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030282; 03-H-0282
Record Dates: First submitted 2003-09-09; First posted 2003-09-09 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hereditary Hemochromatosis
Keywords: Hereditary Disease; Diastolic Dysfunction; Exercise Tolerance; Exercise Stress Echocardiography; MRI; Natural History
MeSH Terms: conditions — Hemochromatosis; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Untreated-NYHA Class I HH subjects without conventional therapy for HH
- 2: Treated- NYHA Class I HH subjects with conventional phlebotomy and/or iron chelation therapy
- 3: Age-gender matched healthy HH control volunteers

SUMMARY:
This study will examine the effect of iron buildup in the hearts of patients with hereditary hemochromatosis (HH), a genetic disease that causes the body to accumulate excess amounts of iron. The excess iron can damage the heart, liver, pancreas, skin, and joints. Generally, early treatment with phlebotomy (periodic removal of a unit of blood), and in some cases chelation (using a drug to remove iron from the body) slows down organ damage in HH patients. This study will try to elucidate the effect of iron buildup in the heart and determine if phlebotomy and chelation help keep the heart healthy.

Patients with HH and healthy volunteers 21 years of age and older may be eligible for this study. (Normal volunteers will provide normal values of heart function that will be used to verify abnormalities detected in HH patients.) Patients must have a gene abnormality of Hfe gene Cys282Try homozygote. They may or may not be receiving treatment for HH and they must have no heart symptoms or serious organ damage due to HH. Candidates will be screened with a medical history and physical examination, blood tests, electrocardiogram (EKG), Holter EKG (24-hour EKG monitoring, see description below), and chest x-ray.

Participants will undergo the following tests and procedures over 2 to 5 days:

* Exercise test: The participant exercises on a treadmill while wearing a mouthpiece, which is used to measure how much oxygen is used. Electrodes placed on the chest and arms monitor the heartbeat during the test.
* Echocardiography: This ultrasound test uses sound waves to take pictures. A small probe is held against the chest to allow a technician to take pictures of the heart and assess its function. A drug called Optison may be injected in an arm vein if needed to enhance the ultrasound images.
* Exercise stress echocardiography: The participant exercises on a stationary bike while heart function is measured with an echocardiogram, EKG, and blood pressure cuff.
* 24-hour Holter EKG: The participant wears a small machine that records heart rhythm continuously for 24 hours. The recorder is connected by cables to electrodes placed on the chest.
* Magnetic resonance imaging: This test uses a magnetic field and radio waves to obtain detailed images of the heart and blood vessels. The participant lies flat on a table that slides inside the scanner, which is a large hollow tube.

All tests are performed once in normal volunteers and in patients who have received standard treatment for HH. Untreated patients repeat the tests 6 months after beginning phlebotomy or chelation. Additional time points for these tests might be added if further evaluation is needed.

DETAILED DESCRIPTION:
Hereditary hemochromatosis (HH) is the most common hereditary metabolic abnormality among Caucasians. Homozygosity for the Cys282Tyr mutation, which is the most common known mutation with a predisposition to iron overload, occurs with an estimated frequency of 8 per 1000 in the Caucasians. Hemochromatosis in its advanced stages is associated with severe cardiac complications including congestive heart failure, premature coronary artery disease, and cardiac arrhythmias. The clinical manifestations of HH are due to increased iron absorption and abnormal iron cycling with excessive iron deposition in various organs. Mutations of the Hfe gene on chromosome 6 have been recently identified. Although the pathophysiology remains incompletely understood, a homozygote mutation in Cys282Tyr is present in 84 to 100% of clinically confirmed HH cases. This discovery permits the early diagnosis of this disease and could be used for screening to identify asymptomatic cases. Therefore, the NHLBI in January 2000 launched a 30 million dollar project named HEIRS (HEmochromatosis and IRon overload Study) to screen 1,000,000 adults for HH, and recently completed enrollment.

<TAB>

Increased left ventricular wall thickness and mass has been found to be early cardiac manifestations of HH appearing before the onset of contractile dysfunction. Interestingly, a report also indicates that functional abnormalities of the heart can be seen in predominantly asymptomatic HH patient group. Such abnormalities of diastolic function are detected by Doppler echocardiography. Observations support the theory that asymptomatic cardiac dysfunction is detectable with non-invasive cardiac imaging in patients with HH. <TAB>

<TAB>

Although the pathophysiology of cardiac dysfunction in HH has not been well characterized, it is speculated that enhanced production of reactive oxygen species (ROS) may be responsible for tissue damage. Therefore, biochemical and/or genetic markers of oxidant stress might be helpful in determining whether this mechanism is involved in producing cardiac dysfunction.

In this protocol, we propose a retrospective pilot study with a small-sized nested prospective study of cardiac function in patients with HH. The intention is to utilize obtained results to design a larger definitive study if results are warranted. The following hypotheses will be tested: Cardiac abnormalities 1) can be diagnosed with conventional non-invasive cardiac imaging in HH patients with New York Heart Association Functional Class I (asymptomatic), 2) limit patients' exercise capacity, 3) are associated with an elevated oxidant stress level, and 4) are improved by phlebotomy and its efficacy correlated with a reduction in oxidant stress.

ELIGIBILITY:
* INCLUSION CRITERIA:

HH Patients

Group A patients (untreated HH patients)

Adults 21 years or older

New York Heart Association Functional Classification Class I

Documented positive phenotyping for homozygote Cys282Tyr of Hfe gene with documented serum ferritin level above 400 ng/ml or documented % iron saturation more than 60%.

Patient has not received standard chronic phlebotomy or deferoxamine treatment. Individuals are allowed to have up to 3 emergency phlebotomies for alleviation of severe iron accumulation before enrollment.

Group B patients (treated HH patients)

Adults 21 years or older

New York Heart Association Functional Classification Class I

Documented positive phenotyping for homozygote Cys282Tyr of Hfe gene with documented serum ferritin level above 400 ng/ml or documented % iron saturation more than 60%.

Patient has been compliant with standard phlebotomy and/or deferoxamine treatment for 6 months or longer and in stable phase with iron saturation 50% or less.

Healthy Volunteers

Group C Patients (Age-Gender Matched Healthy Control Subjects)

Adults 21 years or older.

No symptoms suggestive of heart disease or any other medical conditions, negative Hfe genotyping for Cys282Tyr or His63Asp with normal ferritin and iron saturation.

EXCLUSION CRITERIA:

HH patients

Group A patients (untreated HH patients)

Pregnant or lactating women

History or present evidence of coronary artery disease, heart failure, peripheral vascular disease, coagulopathy, or uncontrolled hypertension (systolic blood pressure over 170 mmHg and/or diastolic pressure over 100 mmHg).

History of significant end-organ damage secondary to HH.

Serum creatinine greater than 2.0 mg/ml

LFT's more than 2.5 times above upper limit of normal

History of structural cardiac disease except mitral valve prolapse with mild mitral regurgitation

Uncontrolled glucose levels with hemoglobin A(1c) above 8 mg/dl or the use of more than one oral hyperglycemic agents or insulin therapy to control diabetes.

Current use of antioxidant treatment such as vitamin E and C. However, the cessation of this treatment 4 weeks prior to the study will allow for inclusion.

Evidence of impaired immunity including HIV

Chronic systemic inflammatory disease such as SLE, rheumatoid arthritis, collagen vascular disease.

Participation in unrelated research involving investigational pharmacological agent in past 30 days.

Current alcohol use (more than 26 grams averaged ethanol intake per day) or drug abuse.

Inability to provide informed consent

Smoking in past 3 months.

Use of beta-adrenergic blocking agents and calcium channel blockers with negative chronotropic effect within 1 week.

Inability to perform treadmill or bicycle exercise testing.

Inability to undergo MRI such as ferromagnetic implant.

Group B patients (treated HH patients)

Pregnant or lactating women

History or present evidence of coronary artery disease, heart failure, peripheral vascular disease, coagulopathy, or uncontrolled hypertension (systolic blood pressure over 170 mmHg and/or diastolic pressure over 100 mmHg).

History of significant end-organ damage secondary to HH.

Serum creatinine greater than 2.0 mg/ml

LFT's more than 2.5 times above upper limit of normal

History of structural cardiac disease except mitral valve prolapse with mild mitral regurgitation

Uncontrolled glucose levels with hemoglobin A(1c) above 8 mg/dl or the use of more than one oral hyperglycemic agents or insulin therapy to control diabetes.

Current use of antioxidant treatment such as vitamin E and C. However, the cessation of this treatment 4 weeks prior to the study will allow for inclusion.

Evidence of impaired immunity including HIV

Chronic systemic inflammatory disease such as SLE, rheumatoid arthritis, collagen vascular disease.

Participation in unrelated research involving investigational pharmacological agent in past 30 days.

Current alcohol use (more than 26 grams averaged ethanol intake per day) or drug abuse.

Inability to provide informed consent

Smoking in past 3 months.

Use of beta-adrenergic blocking agents and calcium channel blockers with negative chronotropic effect within 1 week.

Inability to perform treadmill or bicycle exercise testing.

Inability to undergo MRI such as ferromagnetic implant.

Healthy volunteers

Group C Patients (Age-Gender Matched Healthy Control Subjects)

Pregnant or lactating women.

History or present evidence of any structural cardiac disease except mitral valve prolapse with mild mitral regurgitation, heart failure, peripheral vascular disease, coagulopathy, and uncontrolled hypertension (systolic blood pressure over 170 mmHg and/or diastolic pressure over 100 mmHg).

Serum creatinine greater than 2.0 mg/ml.

LFT's more than 2.5 times above upper limit of normal.

Current use of antioxidant treatment such as vitamin E and C. However, the cessation of this treatment 4 weeks prior to the study will be included.

Uncontrolled glucose levels with hemoglobin A(1C) above 8 mg/dl or the use of oral hyperglycemic agents or insulin therapy to control diabetes.

Evidence of impaired immunity including HIV.

Chronic systemic inflammatory disease such as SLE, rheumatoid arthritis, collagen vascular disease.

Participation in unrelated research involving investigational pharmacological agent in past 30 days.

Current alcohol use (more than 26 grams averaged ethanol intake per day) or drug abuse.

Inability to provide informed consent.

Smoking in past 3 months.

Subjects with any chronic medical problems*

Inability to undergo MRI such as ferromagnetic implant.

*For the purpose of this protocol "chronic medical problems' is defined as any current condition not amenable to curative therapy and which requires long-term medical treatment and/or clinical monitoring.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the North American continent and United States possessions. The patients currently followed at the Transfusion Medicine Department under IRB protocol # 01-CC-0045 will be informed of our study protocol. Also, subjects referred to IRB protocol # 01-CC-0045 from the ongoing genotyping study by the NHLBI (HEIRS trial) will be considered for the potential subjects. Advertisements of our study both on the Web and the NIH newsletters will be planned through the NIH Patient Recruitment and Public Liaison to recruit additional patients if necessary. There will be no exclusion from participation in the study on the basis of ethnicity/race/gender. Since HH is predominantly seen in Caucasian origins and the exact frequency in African, Asian, Hispanic population is too low to estimate, we assume that the study population will not be the same as the demographic representation of ethnic groups in this country because of the inheritance nature of this disease.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2003-12-08 (Actual); Primary Completion 2010-11-12 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Echocardographic variable early diastolic peak tissue Doppler velocity of septal mitral annulus (Em). | 5 year
  To assess detailed cardiac function using non-invasive cardiac imaging in Group A; untreated-NYHA Class I HH subjects without conventional therapy for HH, Group B; treated- NYHA Class I HH subjects with conventional phlebotomy and/or iron chelation therapy and compare these results to those from Group C; age-gender matched healthy control volunteers.
Exercise testing variable change in ejection fraction in response to exercise | 5 year
  To compare the results of the cardiac functional abnormalities in HH to those from healthy control. volunteers. change in ejection fraction in response to exercise (change EF)

CONTACTS AND LOCATIONS:
Overall Officials: My-Le Nguyen, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shizukuda Y, Bolan CD, Tripodi DJ, Yau YY, Nguyen TT, Botello G, Sachdev V, Sidenko S, Ernst I, Waclawiw MA, Leitman SF, Rosing DR. Significance of left atrial contractile function in asymptomatic subjects with hereditary hemochromatosis. Am J Cardiol. 2006 Oct 1;98(7):954-9. doi: 10.1016/j.amjcard.2006.04.040. Epub 2006 Aug 15. PMID 16996882
- [Background] Shizukuda Y, Tripodi DJ, Smith KP, Arena R, Waclawiw MA, Rosing DR. Can we use heart rate recovery information generated by supine ergometry exercise? Am J Cardiol. 2006 Nov 1;98(9):1297-8. doi: 10.1016/j.amjcard.2006.07.009. Epub 2006 Aug 31. No abstract available. PMID 17056351
- [Background] Shizukuda Y, Bolan CD, Tripodi DJ, Yau YY, Smith KP, Sachdev V, Birdsall CW, Sidenko S, Waclawiw MA, Leitman SF, Rosing DR. Left ventricular systolic function during stress echocardiography exercise in subjects with asymptomatic hereditary hemochromatosis. Am J Cardiol. 2006 Sep 1;98(5):694-8. doi: 10.1016/j.amjcard.2006.03.055. Epub 2006 Jul 7. PMID 16923464
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-H-0282.html